CLINICAL TRIAL: NCT04736628
Title: Randomised, Double-blind (Within Dose Groups), Placebo Controlled and Parallel Group Trial to Investigate the Effects of Different Doses of Oral BI 685509 Given Over 20 Weeks on UACR Reduction in Patients With Non-diabetic Kidney Disease
Brief Title: A Study to Test the Effect of Different Doses of Avenciguat (BI 685509) on Kidney Function in People With Chronic Kidney Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1366-0022; 2020-002930-33 (EudraCT Number)
Record Dates: First submitted 2021-02-01; First posted 2021-02-03 (Actual); Results first posted 2024-09-04 (Actual); Last update posted 2024-09-04 (Actual); Status verified 2024-08

CONDITIONS: Chronic Kidney Disease
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Avenciguat 1 mg TID (Experimental): TID=ter in die (3 times a day)
  Interventions: Drug: Avenciguat
- Avenciguat 2 mg TID (Experimental)
  Interventions: Drug: Avenciguat
- Avenciguat 3 mg TID (Experimental)
  Interventions: Drug: Avenciguat
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Avenciguat — Avenciguat
  Other Names: BI 685509
  Arms: Avenciguat 1 mg TID; Avenciguat 2 mg TID; Avenciguat 3 mg TID
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This study is open to adults who have kidney disease that is not caused by diabetes. The purpose of the study is to find out whether a medicine called avenciguat (BI 685509) improves kidney function. Three different doses of avenciguat are tested in this study.

Participants get either one of the three doses of avenciguat or placebo. It is decided by chance who gets which avenciguat dose and who gets placebo. Participants take avenciguat or placebo as tablets 3 times a day. Placebo tablets look like avenciguat tablets but do not contain any medicine. Participants continue taking their usual medicine for kidney disease throughout the study.

Participants are in the study for about 7 months. During this time, they visit the study site about 11 times. Where possible, about 6 of the 11 visits can be done at the participant's home instead of the study site. The trial staff may also contact the participants by phone or video call.

Kidney function is assessed based on the analysis of urine samples, which participants collect at home. At the end of the trial the results are compared between the different doses of avenciguat and placebo. During the study, the doctors also regularly check the general health of the participants.

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated written informed consent in accordance with International Council on Harmonisation-Good Clinical Practice (ICH-GCP) and local legislation prior to admission to the trial.
* Male or female patients aged ≥18 years at time of consent.
* Estimated glomerular filtration rate (eGFR) (Chronic Kidney Disease Epidemiology Collaboration [CKD-EPI] formula) ≥ 20 and < 90 mL/min/1.73 m2 at Visit 1 by central laboratory analysis. eGFR must remain ≥20 mL/min/1.73 m2 after Visit 1 up to the start of Visit 3, measured by central or any local laboratory analysis.
* Urine albumin creatinine ratio (UACR) ≥ 200 and < 3,500 mg/g in spot urine (midstream urine sample) by central laboratory analysis at Visit 1.
* Patients with macroalbuminuria (>300 mg/g) should be treated with the highest tolerated dose of either Angiotensin Converting Enzyme inhibitor (ACEi) or Angiotensin Receptor Blocker (ARB) (but not both). For patients with microalbuminuria the use of ACEi or ARB is at the discretion of the Investigator. Treatment should be at a stable dose for ≥ 4 weeks before Visit 1 with no planned change of the therapy during the trial.
* If the patient is taking any of the following medications they should be on a stable dose at least 4 weeks prior to visit 1 until start of treatment, with no planned change of the therapy during the trial: anti-hypertensives, non-steroidal anti-inflammatory drugs (NSAIDs), endothelin receptor antagonists, systemic steroids or Sodium-glucose co-transporter-2 (SGLT2) inhibitors.
* In the Investigator's judgment any kind of diagnosed chronic kidney disease whose primary cause is clinically not considered to be of diabetic origin.

Further inclusion criteria apply

Exclusion Criteria:

* Treatment with Renin Angiotensin Aldosterone System (RAAS) interventions (apart from either ACEi or ARB), Phosphodiesterase-5-inhibitors, non-specific phosphodiesterase inhibitors (such as dipyridamole and theophylline), Nitric Oxide (NO) donors including nitrates, soluble Guanylate Cyclase (sGC)-stimulators/activators (other than trial treatment) or any other restricted medication (including Organic Anion-Transporting Polypeptide 1B1 and 1B3 (OATP1B1/3) inhibitors, Uridine 5'-diphosphate -glucuronosyltransferase (UGT) inhibitors/inducers) as provided in the Investigator Site File (ISF) within 4 weeks prior to visit 1 and throughout screening and baseline run-in. Patients who must or wish to continue the intake of restricted medications or any drug considered likely to interfere with the safe conduct of the trial.
* Any clinically relevant laboratory value from screening until start of trial treatment which, in the investigator's judgement, puts the patient at additional risk.
* Diagnosed with diabetic kidney disease.
* Any immunosuppression therapy or immunotherapy in last 3 months prior to visit 1 and throughout screening and baseline run-in (except prednisolone ≤10 mg or equivalent).
* Acute kidney injury (AKI) according to the Kidney Disease: Improving Global Outcomes (KDIGO) definition in the 30 days prior to Visit 1 until the start of trial treatment.
* Planned start of chronic renal replacement therapy during the trial or end stage renal disease before start of trial treatment.
* Known history of moderate or severe symptomatic orthostatic dysregulation as judged by the investigator before start of trial treatment.
* The patient has an active infection with Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2) (or is known to have a positive test from screening until randomisation).
* Further exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 261 (Actual)
Dates: Start 2021-04-27 (Actual); Primary Completion 2023-08-15 (Actual); Study Completion 2023-09-21 (Actual)

CONTACTS AND LOCATIONS:
Locations (110):
- United States (23):
  - Clearview Medical Research, LLC, Canyon Country, California
  - Rancho Cucamonga Clinical Trials, Rancho Cucamonga, California
  - Kidney & Hypertension Center, Victorville, California
  - Chase Medical Research, LLC, Waterbury, Connecticut
  - Nephrology Associates, P.A., Newark, Delaware
  - Indago Research and Health Center, Hialeah, Florida
  - Homestead Associates in Research, Miami, Florida
  - Bioclinical Research Alliance, Inc., Miami, Florida
  - Alma Clinical Research, Inc., Miami, Florida
  - Panax Clinical Research, Miami Lakes, Florida
  - Davita Clinical Research, Columbus, Georgia
  - Meridian Clinical Research, LLC, Savannah, Georgia
  - Boise Kidney and Hypertension, PLLC, Boise, Idaho
  - Research by Design, LLC, Chicago, Illinois
  - Renal Associates of Baton Rouge, Baton Rouge, Louisiana
  - DaVita Clinical Research, Las Vegas, Nevada
  - Nevada Kidney Disease and Hypertension Centers, PLLC, Las Vegas, Nevada
  - New Jersey Kidney Care, LLC, Jersey City, New Jersey
  - Brookview Hills Research Associates LLC, Winston-Salem, North Carolina
  - Knoxville Kidney Center PLLC, Knoxville, Tennessee
  - Davita Clinical Research, El Paso, Texas
  - Clinical Advancement Center, PLLC, San Antonio, Texas
  - Kidney Specialists of North Houston, PLLC, Shenandoah, Texas
- Argentina (9):
  - STAT Research, CABA
  - CEDIC - Centro de Investigacion Clinica, CABA
  - CEMIC, CABA
  - Instituto Privado de Investigaciones Clínica Córdoba S.A., Córdoba
  - Centro de Investigaciones Médicas Mar del Plata, Mar del Plata
  - Instituto de Investigaciones Clinicas Mar del Plata, Mar del Plata
  - Instituto Médico Catamarca - IMEC, Rosario
  - CEDIR Santa Fe, Santa Fe
  - CEREHA S.A.- Centro de Estudios Renales e Hipertensión Arterial, Sarandí
- Australia (7):
  - Renal Research, Gosford, Gosford, New South Wales
  - Nepean Hospital, Kingswood, New South Wales
  - Macquarie University, Macquarie Park, New South Wales
  - Royal North Shore Hospital, St Leonards, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Austin Health, Heidelberg, Victoria
  - Royal Melbourne Hospital, Parkville, Victoria
- Canada (5):
  - CARe Clinic, Red Deer, Alberta
  - Stouffville Medical Centre, Stouffville, Ontario
  - Toronto General Hospital, Toronto, Ontario
  - Albion Finch Medical Centre, Toronto, Ontario
  - Fadia El Boreky Medicine Professional, Waterloo, Ontario
- China (6):
  - Peking University First Hospital, Beijing
  - Peking University People's Hospital, Beijing
  - Peking University Third Hospital, Beijing
  - People's Hospital of Sichuan Province, Chengdu
  - Second Affiliated Hospital Chongqing Medical University, Chongqing
  - The People's Hospital Of Xuancheng City, Xuancheng
- Denmark (4):
  - Aarhus University Hospital, Aarhus N
  - Herlev and Gentofte Hospital, Herlev
  - Holbæk Sygehus, Holbæk
  - Sjællands Universitetshospital, Roskilde
- Germany (2):
  - Klinikum Region Hannover GmbH, Hanover
  - Universitätsklinikum Schleswig-Holstein, Campus Lübeck, Lübeck
- Hong Kong (4):
  - Prince of Wales Hospital, Hong Kong
  - Princess Margaret Hospital, Hong Kong
  - Queen Mary Hospital, Hong Kong
  - Tung Wah Hospital, Hong Kong
- Japan (15):
  - Chubu Rosai Hospital, Aichi, Nagoya
  - Daido Hospital, Aichi, Nagoya
  - Juntendo University Urayasu Hospital, Chiba, Urayasu
  - Kurume University Hospital, Fukuoka, Kurume
  - Nakayamadera Imai Clinic, Hyogo, Takarazuka
  - Takai Naika Clinic, Kanagawa, Kamakura
  - Kyoto University Hospital, Kyoto, Kyoto
  - Kuana City Medical Center, Mie, Kuwana
  - Shinshu University Hospital, Nagano, Matsumoto
  - Kawasaki Medical School Hospital, Okayama, Kurashiki
  - Saitama Medical University Hospital, Saitama, Iruma-gun
  - Yaizu City Hospital, Shizuoka, Yaizu
  - The University of Tokyo Hospital, Tokyo, Bunkyo-ku
  - Tokyo-Eki Center-building Clinic, Tokyo, Chuo-ku
  - Nihon University Itabashi Hospital, Tokyo, Itabashi-ku
- Malaysia (5):
  - University Kebangsaan Malaysia, Cheras, Kuala Lumpur
  - Hospital Raja Permaisuri Bainun, Ipoh, Perak
  - Universiti Sains Malaysia Hospital, Kelantan
  - University of Malaya Medical Centre, Kuala Lumpur
  - Hospital Selayang, Kuala Selangor
- Mexico (6):
  - Centro de Investigacion Cardiometabolica de Aguascalientes, Aguascalientes
  - Centenario Hospital Miguel Hidalgo, Aguascalientes
  - Instituto Nacional de Cs Médicas y Nutrición S Zubiran, Mexico City
  - Instituto Nacional de Cardiologia Ignacio Chavez, Mexico City
  - Clinstile S.A. de C.V., México
  - Hospital Universitario Dr Jose Eleuterio Gonzalez, Monterrey
- New Zealand (3):
  - Dunedin Hospital, Dunedin
  - P3 Research Kapiti, Paraparaumu
  - P3 Research, Tauranga
- Poland (4):
  - Cardiovascular Centre of Malopolska, Chrzanów
  - Pratia MCM Krakow, Krakow
  - Cent.Clin.Hosp.Med.Univ.Lodz, Lodz
  - Medicome Limited Liability Company, Oświęcim
- Portugal (4):
  - ULS da Região de Aveiro, Aveiro
  - CHLO, EPE - Hospital de Santa Cruz, Carnaxide
  - ULS de Santa Maria, E.P.E, Lisbon
  - Centro Hospitalar Universitário São João,EPE, Porto
- Russia (2):
  - Moscow 1st State Med.Univ.n.a.I.M.Sechenov, Moscow
  - St. Petersburg GUZ City Hospital no. 31, St. Petersburg, Saint Petersburg
- Spain (7):
  - Hospital Vall d'Hebron, Barcelona
  - Hospital de Bellvitge, L'Hospitalet de Llobregat
  - Fundación Jiménez Díaz, Madrid
  - Clínica Universidad de Navarra, Pamplona
  - Hospital Virgen Macarena, Seville
  - Hospital Clínico de Valencia, Valencia
  - Hospital Dr. Peset, Valencia
- ProbarE i Stockholm, Stockholm, Sweden
- United Kingdom (3):
  - Lakeside Surgery, Corby
  - University Hospital Coventry, Coventry
  - Barts and The London School of Medicine and Dentistry, London

IPD SHARING:
Plan to Share IPD: Yes
After the study is completed and the primary manuscript is accepted for publishing, researchers can use this following link https://www.mystudywindow.com/msw/datasharing to request access to the clinical study documents regarding this study, and upon a signed "Document Sharing Agreement". Also, Researchers can use the following link https://www.mystudywindow.com/msw/datasharing to find information in order to request access to the clinical study data, for this and other listed studies, after the submission of a research proposal and according to the terms outlined in the website.
  The data shared are the raw clinical study data sets.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: After all regulatory activities are completed in the US and EU for the product and indication, and after the primary manuscript has been accepted for publication.
Access Criteria: For study documents - upon signing of a 'Document Sharing Agreement'. For study data - 1. after the submission and approval of the research proposal (checks will be performed by both the independent review panel and the sponsor, including checking that the planned analysis does not compete with sponsor's publication plan); 2. and upon signing of a 'Data Sharing Agreement'.
URL: https://www.mystudywindow.com/msw/datasharing

REFERENCES:
- [Derived] Heerspink HJL, Cherney D, Gafor AHA, Gorriz JL, Pergola PE, Tang SCW, Desch M, Iliev H, Sun Z, Steubl D, Nangaku M. Effect of Avenciguat on Albuminuria in Patients with CKD: Two Randomized Placebo-Controlled Trials. J Am Soc Nephrol. 2024 Sep 1;35(9):1227-1239. doi: 10.1681/ASN.0000000000000418. Epub 2024 May 25. PMID 38795055
- See also: Related Info — https://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This trial was a Phase II, randomised, placebo-controlled, double-blind (within dose groups), parallel, multicentre clinical trial in patients with non-diabetic kidney disease (non-DKD) to demonstrate the effectiveness and safety of avenciguat and to characterize the dose-response relationship for avenciguat in patients with non-DKD by assessing 3 doses and placebo.
Pre-assignment Details: Patients underwent a screening period of up to 3 weeks from the time of informed consent. After confirmation of eligibility at screening, patients continued in a 2-week baseline run-in period. Patients who successfully completed the screening and baseline run-in periods and met the inclusion/exclusion criteria were randomised equally into 1 of 3 parallel dose groups, and in each dose group to treatment either with avenciguat or matching placebo in a 3:1 ratio.
Groups:
- Avenciguat 1 mg TID: Patients received daily orally one film-coated tablet of 1 milligram (mg) of avenciguat three times a day (TID) in Weeks 1 to 20 (included).
  Avenciguat had to be taken with a glass of water and could be taken with or without food.
  Patients continued the treatment until undue drug toxicity, disease progression, or withdrawal of consent, whichever occurred first.
- Avenciguat 2 mg TID: Patients received daily orally one film-coated tablet of 1 milligram (mg) of avenciguat three times a day (TID) in Week 1 and Week 2. If the 1 mg TID medication was tolerated, up-titration to 2 mg of avenciguat (one film-coated tablet of 2 mg) TID occurred after 2 weeks until Week 20 of treatment.
  Avenciguat had to be taken with a glass of water and could be taken with or without food.
  Patients continued the treatment until undue drug toxicity, disease progression, or withdrawal of consent, whichever occurred first.
- Avenciguat 3 mg TID: Patients received daily orally one film-coated tablet of 1 milligram (mg) of avenciguat three times a day (TID) in Week 1 and Week 2. If the 1 mg TID medication was tolerated, up-titration to 2 mg avenciguat (one film-coated tablet of 2 mg) TID occurred after 2 weeks until Week 4 of treatment. Then if medication was tolerated, up-titration to 3 mg avenciguat (one film-coated tablet of 3 mg) TID occurred from Week 5 until Week 20.
  Avenciguat had to be taken with a glass of water and could be taken with or without food.
  Patients continued the treatment until undue drug toxicity, disease progression, or withdrawal of consent, whichever occurred first.
- Placebo: This arm comprises all placebo treated participants. Participants were administered film-coated tablets of placebo matching avenciguat 1mg, 2mg or 3mg 3 times a day (TID) during 20 weeks of treatment.
  Placebo matching avenciguat had to be taken with a glass of water and could be taken with or without food.
  Patients continued the treatment until undue drug toxicity, disease progression, or withdrawal of consent, whichever occurred first.
Period: Overall Study
Arm/Group | Avenciguat 1 mg TID | Avenciguat 2 mg TID | Avenciguat 3 mg TID | Placebo
Started (Randomised to avenciguat or placebo matching avenciguat) | 64 | 65 | 66 | 66
Treated | 64 | 65 | 66 | 64
Completed | 58 | 60 | 60 | 55
Not Completed | 6 | 5 | 6 | 11
Not completed — Not treated | 0 | 0 | 0 | 2
Not completed — Other reason than listed | 1 | 2 | 2 | 3
Not completed — Protocol deviation | 0 | 0 | 0 | 1
Not completed — Burden of study procedures | 1 | 0 | 0 | 1
Not completed — Change of residence | 0 | 1 | 0 | 0
Not completed — Perceived lack of efficacy | 1 | 0 | 0 | 1
Not completed — Adverse Event | 3 | 2 | 4 | 3

BASELINE CHARACTERISTICS:
Population: Randomised Set (RS): this patient set included all entered and randomised patients.
Groups:
- Total: Total of all reporting groups
Arm/Group | Avenciguat 1 mg TID | Avenciguat 2 mg TID | Avenciguat 3 mg TID | Placebo | Total
Number analyzed (Participants) | 64 | 65 | 66 | 66 | 261
Age, Continuous [Mean (Standard Deviation); unit: Years] | 54.6 (16.3) | 60.4 (15.5) | 59.3 (15.0) | 58.1 (14.4) | 58.1 (15.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 16 | 26 | 17 | 80
  Male | 43 | 49 | 40 | 49 | 181
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 18 | 20 | 11 | 18 | 67
  Not Hispanic or Latino | 46 | 45 | 55 | 48 | 194
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 4 | 1 | 4 | 12
  Asian | 18 | 20 | 12 | 15 | 65
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 2 | 1 | 3
  Black or African American | 3 | 1 | 8 | 5 | 17
  White | 39 | 38 | 42 | 40 | 159
  More than one race | 1 | 1 | 0 | 0 | 2
  Unknown or Not Reported | 0 | 1 | 1 | 1 | 3
Sodium-glucose cotransporter 2 inhibitor (SGLT2i) use at randomization [Count of Participants; unit: Participants] — Number of patients in each category sodium-glucose cotransporter 2 inhibitor (SGLT2i) use at randomization. The reported categories of SGLT2i use at randomization are: Yes; No.
  Participants
    Yes | 17 | 14 | 15 | 16 | 62
    No | 47 | 51 | 51 | 50 | 199
Baseline urine albumine creatinine ratio (UACR), 10-hour urine [Mean (Standard Deviation); unit: milligram/gram] — Baseline UACR measured in 10-hour urine is reported. UACR is a ratio between two measured substances i.e., albumine and creatinine and it is calculated as: (Urine albumin (milligram (mg)/deciliter (dL)))/(urine creatinine gram (g)/deciliter (dL))= UACR in mg/g. Albuminuria is present when UACR is greater than 30 mg/g and is a marker for chronic kidney disease (CKD). Baseline was defined as the mean of all non-missing assessments from visit 2 (Week -2) until prior to the first intake of trial medication.
  milligram/gram | 1024.1 (920.1) | 868.2 (727.7) | 941.5 (1155.2) | 1076.2 (1786.2) | 977.6 (1213.7)
Baseline Urine Albumine Creatinine Ratio (UACR) in First Morning Void (FMV) [Mean (Standard Deviation); unit: milligram/gram] — UACR measured in FMV is reported. UACR is a ratio between two measured substances i.e., albumine and creatinine and it is calculated as: (urine albumin (milligram (mg)/deciliter (dL)))/(urine creatinine gram (g)/deciliter (dL))= UACR in mg/g. Albuminuria is present when UACR is greater than 30 mg/g and is a marker for chronic kidney disease (CKD). Baseline was defined as the mean of all non-missing assessments from visit 2 (Week -2) until prior to the first intake of trial medication.
  milligram/gram | 879.1 (840.8) | 745.4 (661.9) | 821.3 (1083.5) | 874.1 (1142.0) | 829.9 (949.5)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Log Transformed Urine Albumin Creatinine Ratio (UACR) Measured in 10-hour Urine After 20 Weeks of Trial Treatment
Description: Change from baseline in log transformed Urine Albumin Creatinine Ratio (UACR) measured in 10-hour urine after 20 weeks of trial treatment is reported.
  Least Squares Mean (Standard error) were estimated by restricted maximum likelihood (REML)-based mixed-effect model for repeated measures (MMRM) including the fixed, categorical effects of treatment at each visit (baseline, Week 6, Week 12, and Week 20), and the continuous effect of baseline at each visit (Week 6, Week 12, and Week 20) as well as random effects of patient.
  Log transformed UACR at Week 20 was log of (average of all available scheduled measurements between week 18 and week 20).
  The data in the Outcome Measure Data Table represent the Least Squares Mean (Standard error) at Week 20.
Time Frame: The MMRM model is a longitudinal analysis and it incorporated UACR measurements from baseline (Week -2, Week -1, Week 0 pre-dose) and Week 6, Week 12 and Week 20. The data represent the Least Squares Mean at Week 20.
Population: Full Analysis Set (FAS): included all patients who had at least one baseline measurement of UACR in Week -2, -1, or 0 and at least 1 post-baseline measurement after Week 6.
Measure: Least Squares Mean (Standard Error); unit: log (mg/g)
Arm/Group | Avenciguat 1 mg TID | Avenciguat 2 mg TID | Avenciguat 3 mg TID | Placebo
Number analyzed (Participants) | 64 | 61 | 62 | 62
log (mg/g) | -0.210 (0.067) | -0.190 (0.068) | -0.217 (0.068) | 0.018 (0.068)
Statistical Analysis 1: Comparison: Avenciguat 1 mg TID vs Placebo; Least Squares Mean differences and 95% confidence intervals were estimated by restricted maximum likelihood (REML)-based mixed-effect model for repeated measures (MMRM) including the fixed, categorical effects of treatment at each visit (baseline, Week 6, Week 12 and Week 20), and the continuous effect of baseline at each visit (Week 6, Week 12, and Week 20) as well as random effects of patient; Test type: Other; p = 0.0179, Mixed-effect Model repeat Measurement; Mean Difference (Net) = -0.228, 95% CI 2-sided [-0.417 to -0.040] — Least Squares Mean of "Avenciguat 1 mg TID" - Least Squares Mean of "Placebo"
Statistical Analysis 2: Comparison: Avenciguat 2 mg TID vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.0307, Mixed-effect Model repeat Measurement; Mean Difference (Net) = -0.209, 95% CI 2-sided [-0.398 to -0.020] — Least Squares Mean of "Avenciguat 2 mg TID" - Least Squares Mean of "Placebo"
Statistical Analysis 3: Comparison: Avenciguat 3 mg TID vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.0151, Mixed-effect Model repeat Measurement; Mean Difference (Net) = -0.235, 95% CI 2-sided [-0.425 to -0.046] — Least Squares Mean of "Avenciguat 3 mg TID" - Least Squares Mean of "Placebo"
Statistical Analysis 4: Comparison: Avenciguat 1 mg TID vs Avenciguat 2 mg TID vs Avenciguat 3 mg TID vs Placebo; A flat vs. non-flat dose-response relationship across the 3 doses of avenciguat and placebo was tested using the Multiple Comparison Procedure - Modelling (MCP-Mod) approach which evaluated simultaneously 5 different plausible dose-response patterns (Emax, exponential, linear, quadratic, sigmoid emax) while protecting the overall probability of type I error (one-sided alpha of 0.050). The total daily dose was considered for MCP-Mod analysis (placebo, active avenciguat 3 mg, 6 mg, and 9 mg); Test type: Other — MMRM estimates were used as input for the MCP-Mod. MMRM included the fixed, categorical effects of treatment at each visit (baseline, Week 6, Week 12 and Week 20), and the continuous effect of baseline at each visit (Week 6, Week 12, and Week 20) as well as random effects of patient; p = 0.0053, MCP-Mod E-max model fit; Model assumption: 80% of the maximum effect is achieved at 6 mg
Statistical Analysis 5: Comparison: Avenciguat 1 mg TID vs Avenciguat 2 mg TID vs Avenciguat 3 mg TID vs Placebo; [analysis description as in outcome 1, analysis 4]; Test type: Other — [test comment as in outcome 1, analysis 4]; p = 0.0102, MCP-Mod quadratic model fit; Model assumption: 50 % of the maximum effect is achieved at a dose of 3 mg. 90 % of the maximum effect is achieved at a dose of 6 mg
Statistical Analysis 6: Comparison: Avenciguat 1 mg TID vs Avenciguat 2 mg TID vs Avenciguat 3 mg TID vs Placebo; [analysis description as in outcome 1, analysis 4]; Test type: Other — [test comment as in outcome 1, analysis 4]; p = 0.0230, MCP-Mod linear model fit; Model assumption: no assumption is needed
Statistical Analysis 7: Comparison: Avenciguat 1 mg TID vs Avenciguat 2 mg TID vs Avenciguat 3 mg TID vs Placebo; [analysis description as in outcome 1, analysis 4]; Test type: Other — [test comment as in outcome 1, analysis 4]; p = 0.0292, MCP-Mod Sigmoid Emax model fit; Model assumption: 30 % of the maximum effect is achieved at a dose of 3 mg. 90 % of the maximum effect is achieved at a dose of 6 mg
Statistical Analysis 8: Comparison: Avenciguat 1 mg TID vs Avenciguat 2 mg TID vs Avenciguat 3 mg TID vs Placebo; [analysis description as in outcome 1, analysis 4]; Test type: Other — [test comment as in outcome 1, analysis 4]; p = 0.0468, MCP-Mod Exponential model fit; Model assumption: 20% of the maximum effect is achieved at 3 mg

2. Secondary Outcome: Change From Baseline in Log Transformed UACR Measured in First Morning Void Urine After 20 Weeks of Trial Treatment
Description: Change from baseline in log transformed UACR measured in First Morning Void urine after 20 weeks of trial treatment is reported.
  Least Squares Mean (Standard error) were estimated by restricted maximum likelihood (REML)-based mixed-effect model for repeated measures (MMRM) including the fixed, categorical effects of treatment at each visit (baseline, Week 6, Week 12 and Week 20), and the continuous effect of baseline at each visit (Week 6, Week 12, and Week 20) as well as random effects of patient.
  The first morning void (FMV) was the first urination after the patient woke up at their usual time to start their day. Log transformed UACR at Week 20 was log of (average of all available scheduled measurements between week 18 and week 20). The data in the Outcome Measure Data Table represent the Least Squares Mean (Standard error) at Week 20.
Time Frame: The MMRM model is a longitudinal analysis and it incorporated UACR measurements from baseline (Week -2 and Week -1) and Week 6, Week 12 and Week 20. The data represent the Least Squares Mean at Week 20.
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: log (mg/g)
Arm/Group | Avenciguat 1 mg TID | Avenciguat 2 mg TID | Avenciguat 3 mg TID | Placebo
Number analyzed (Participants) | 64 | 61 | 62 | 62
log (mg/g) | -0.190 (0.071) | -0.180 (0.073) | -0.161 (0.071) | 0.027 (0.072)
Statistical Analysis 1: Comparison: Avenciguat 1 mg TID vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.0327, Mixed-effect Model repeat Measurement; Mean Difference (Net) = -0.217, 95% CI 2-sided [-0.416 to -0.018] — Least Squares Mean of "Avenciguat 1 mg TID" - Least Squares Mean of "Placebo"
Statistical Analysis 2: Comparison: Avenciguat 2 mg TID vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.0447, Mixed-effect Model repeat Measurement; Mean Difference (Net) = -0.206, 95% CI 2-sided [-0.408 to -0.005] — Least Squares Mean of "Avenciguat 2 mg TID" - Least Squares Mean of "Placebo"
Statistical Analysis 3: Comparison: Avenciguat 3 mg TID vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.0654, Mixed-effect Model repeat Measurement; Mean Difference (Net) = -0.187, 95% CI 2-sided [-0.387 to 0.012] — Least Squares Mean of "Avenciguat 3 mg TID" - Least Squares Mean of "Placebo"

3. Secondary Outcome: Number of Patients Achieving UACR Decreases in 10-hour Urine of at Least 20% From Baseline After 20 Weeks of Trial Treatment
Description: Number of patients achieving urine albumin creatinine ratio (UACR) decreases in 10-hour urine of at least 20% from baseline after 20 weeks of trial treatment.
  During the 10-hour period every time the patient urinates, and the patient collected their urine into a provided container. An aliquot of this urine was taken and used as the 10-hour UACR sample.
Time Frame: At baseline (Day -14 and Day -7) and at Week 20 (Day 141) after start of trial treatment.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Avenciguat 1 mg TID | Avenciguat 2 mg TID | Avenciguat 3 mg TID | Placebo
Number analyzed (Participants) | 64 | 61 | 62 | 62
Participants | 25 | 27 | 31 | 14
Statistical Analysis 1: Comparison: Avenciguat 1 mg TID vs Placebo; Treatment and sodium-glucose co-transporter-2 inhibitor (SGLT2i) use at randomization were used as covariates in the logistic regression model; Test type: Other; p = 0.0476, Regression, Logistic — Nominal p-value; Odds Ratio (OR) = 2.20, 95% CI 2-sided [1.01 to 4.79] — Odds ratio (Avenciguat 1 mg TID vs. Placebo)
Statistical Analysis 2: Comparison: Avenciguat 2 mg TID vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Other; p = 0.0119, Regression, Logistic — Nominal p-value; Odds Ratio (OR) = 2.72, 95% CI 2-sided [1.25 to 5.94] — Odds ratio (Avenciguat 2 mg TID vs. Placebo)
Statistical Analysis 3: Comparison: Avenciguat 3 mg TID vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Other; p = 0.0019, Regression, Logistic — Nominal p-value; Odds Ratio (OR) = 3.43, 95% CI 2-sided [1.58 to 7.45] — Odds ratio (Avenciguat 3 mg TID vs. Placebo)

4. Secondary Outcome: Number of Patients Achieving UACR Decreases in First Morning Void Urine of at Least 20% From Baseline After 20 Weeks of Trial Treatment
Description: Number of patients achieving urine albumin creatinine ratio (UACR) decreases in First Morning Void urine of at least 20% from baseline after 20 weeks of trial treatment is reported. The first morning void (FMV) was the first urination after the patient woke up at their usual time to start their day.
Time Frame: At baseline (Day -14 and Day -7) and at Week 20 (Day 141) after start of trial treatment.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Avenciguat 1 mg TID | Avenciguat 2 mg TID | Avenciguat 3 mg TID | Placebo
Number analyzed (Participants) | 64 | 61 | 62 | 62
Participants | 27 | 26 | 26 | 16
Statistical Analysis 1: Comparison: Avenciguat 1 mg TID vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Other; p = 0.0497, Regression, Logistic — Nominal p-value; Odds Ratio (OR) = 2.13, 95% CI 2-sided [1.00 to 4.55] — Odds ratio (Avenciguat 1 mg TID vs. Placebo)
Statistical Analysis 2: Comparison: Avenciguat 2 mg TID vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Other; p = 0.0502, Regression, Logistic — Nominal p-value; Odds Ratio (OR) = 2.15, 95% CI 2-sided [1.00 to 4.61] — Odds ratio (Avenciguat 2 mg TID vs. Placebo)
Statistical Analysis 3: Comparison: Avenciguat 3 mg TID vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Other; p = 0.0572, Regression, Logistic — Nominal p-value; Odds Ratio (OR) = 2.09, 95% CI 2-sided [0.98 to 4.49] — Odds ratio (Avenciguat 3 mg TID vs. Placebo)

ADVERSE EVENTS:
Time Frame: "All-Cause Mortality" "Serious Adverse Events" and "Other Adverse Events": From first avenciguat intake until last avenciguat intake or patient's trial termination date, whichever occurs earlier + 7 days of Residual effect period (REP), up to 148 days.
Description: Treated Set (TS): this patient set included all patients who received at least 1 dose of trial medication.
Arm/Group | Avenciguat 1 mg TID | Avenciguat 2 mg TID | Avenciguat 3 mg TID | Placebo
All-Cause Mortality (participants affected / at risk) | 0/64 | 0/65 | 0/66 | 0/64
Serious Adverse Events (participants affected / at risk) | 3/64 | 3/65 | 6/66 | 6/64
Other Adverse Events (participants affected / at risk) | 17/64 | 19/65 | 26/66 | 21/64
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Avenciguat 1 mg TID (N=64) | Avenciguat 2 mg TID (N=65) | Avenciguat 3 mg TID (N=66) | Placebo (N=64)
Haemorrhagic diathesis (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 1 | 0
Angina pectoris (Cardiac disorders) | 0 | 0 | 1 | 0
Cardiac failure (Cardiac disorders) | 1 | 0 | 0 | 1
Appendicitis noninfective (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Enteritis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 1 | 0
COVID-19 (Infections and infestations) | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1
Pyelonephritis acute (Infections and infestations) | 0 | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Incision site haemorrhage (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 1 | 0
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 2
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Hypertensive urgency (Vascular disorders) | 0 | 0 | 1 | 0
Hypotension (Vascular disorders) | 1 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Avenciguat 1 mg TID (N=64) | Avenciguat 2 mg TID (N=65) | Avenciguat 3 mg TID (N=66) | Placebo (N=64)
Diarrhoea (Gastrointestinal disorders) | 2 | 3 | 6 | 4
Nausea (Gastrointestinal disorders) | 2 | 0 | 4 | 1
Fatigue (General disorders) | 0 | 2 | 6 | 2
Oedema peripheral (General disorders) | 0 | 4 | 5 | 5
COVID-19 (Infections and infestations) | 4 | 5 | 3 | 4
Nasopharyngitis (Infections and infestations) | 4 | 2 | 3 | 2
Gout (Metabolism and nutrition disorders) | 1 | 3 | 5 | 0
Headache (Nervous system disorders) | 5 | 1 | 5 | 3
Hypotension (Vascular disorders) | 3 | 6 | 5 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2022-03-15): https://cdn.clinicaltrials.gov/large-docs/28/NCT04736628/Prot_000.pdf
  • Statistical Analysis Plan (2023-11-01): https://cdn.clinicaltrials.gov/large-docs/28/NCT04736628/SAP_001.pdf